CLINICAL TRIAL: NCT00702104
Title: PSA Screening of African-American Men in The San Francisco Area
Brief Title: Frequency of Prostate-Specific Antigen Screening in African American Men in the San Francisco Area
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000596996; UCSF-0555105; UCSF-H7056-21713-06
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: survey administration

SUMMARY:
RATIONALE: Screening may help doctors find prostate cancer sooner, when it may be easier to treat.

PURPOSE: This research study is looking at whether patients who are being screened for prostate cancer have been previously screened.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the degree to which patients who are being screened for prostate cancer have been previously screened.

OUTLINE: Participants complete questions on a survey about prior prostate-specific antigen blood tests done for the purpose of screening for prostate cancer and are asked about their pastor, church, and how they heard about the SELECT study to determine the degree to which African-American men in a church-going population have been previously screened.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets all of the following criteria:

  * African-American male
  * Age 35 years or older
  * Attends church on a regular basis
  * Resides in the San Francisco area

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Dates: Start 2003-01; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Degree to which patients who are being screened for prostate cancer have been previously screened

CONTACTS AND LOCATIONS:
Overall Officials: Mack Roach, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States